CLINICAL TRIAL: NCT00945815
Title: S0910, A Phase II Study of Epratuzumab (NSC-716711) in Combination With Cytarabine and Clofarabine for Patients With Relapsed or Refractory Ph- Negative Precursor B-Cell Acute Lymphoblastic Leukemia
Brief Title: S0910 Epratuzumab, Cytarabine, and Clofarabine in Treating Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0910; S0910 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Results first posted 2014-01-03 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Leukemia
Keywords: B-cell adult acute lymphoblastic leukemia; L1 adult acute lymphoblastic leukemia; L2 adult acute lymphoblastic leukemia; recurrent adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — epratuzumab; Clofarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): AraC 1 g/m2/d IV Days 1-5 clofarabine 40 mg/m2/d IV Days 2-6 epratuzumab 360 mg/m2/d IV Days 7, 14, 21, 28 acetaminophen 650 mg/d PO Days 7, 14, 21, 28 diphenhydramine 50 mg/d IV Days 7, 14, 21, 28 IT methotrexate 12 mg IT at least 1 wk apart during induction All give 1 cycle
  Interventions: Biological: epratuzumab; Drug: clofarabine; Drug: cytarabine; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: epratuzumab
Drug: clofarabine
Drug: cytarabine
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Monoclonal antibodies, such as epratuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cytarabine and clofarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving epratuzumab together with cytarabine and clofarabine may kill more cancer cells.

PURPOSE: This phase II trial is studying the side effects and how well giving epratuzumab together with cytarabine and clofarabine works in treating patients with relapsed or refractory acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test whether the complete remission (CR) rate (CR and incomplete CR) in adult patients with relapsed or refractory precursor B-cell acute lymphoblastic leukemia is sufficiently high after treatment with cytarabine, clofarabine, and epratuzumab to warrant further investigation.
* To estimate the frequency and severity of toxicities associated with the dosing schedule of cytarabine, clofarabine, and epratuzumab used in this study.
* To investigate, preliminarily, the effect of laboratory correlates (minimal post-treatment residual disease) and cytogenetic factors on prognosis in this patient population. (Not reported here due to limited MRD data)

OUTLINE: This is a multicenter study.

Patients receive cytarabine IV over 2 hours on days 1-5, clofarabine IV over 1 hour on days 2-6, and epratuzumab IV over at least 1 hour on days 7, 14, 21, and 28 in the absence of disease progression or unacceptable toxicity*.

NOTE: * Prophylactic intrathecal methotrexate is required for patients < 22 years of age, and is recommended (but not required) for patients ≥ 22 years of age.

Blood samples, bone marrow samples, and/or tumor tissue samples may be collected for further laboratory analysis.

Patients are followed up every 3 months for 2 years, then annually for 3 years (until 5 years after registration).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Morphologically confirmed precursor B-cell acute lymphoblastic leukemia (ALL) (non T-cell)

  * Must have evidence of disease in bone marrow or peripheral blood

    * Immunophenotyping of the blood or marrow lymphoblasts must be performed to determine lineage (B cell, T cell, or mixed B/T cell)
    * Must have ≥ 5% lymphoblasts present in the blood or bone marrow
    * At least 20% of marrow and/or peripheral blood lymphoblasts must be CD22+ by flow cytometry

      * Co-expression of myeloid antigens (CD13 and CD33) allowed
    * Patients with only extramedullary disease in the absence of bone marrow or blood involvement are not eligible
* Philadelphia (Ph) chromosome-negative disease

  * Patients with unknown Ph status by cytogenetics or FISH and unknown BCR/ABL status by PCR are eligible for study registration, but must be removed from study therapy if found to be Ph+ or BCR/ABL+ after study registration
* Refractory to a standard induction regimen that included vincristine and prednisone or high-dose cytarabine or mitoxantrone OR relapsed after successful prior induction therapy

  * Any number of prior induction therapies or any number of remissions achieved are allowed
* No M0 acute myeloid leukemia, mixed lineage leukemia, or L3 (Burkitt) leukemia
* No active CNS involvement by clinical evaluation

  * Patients with a documented history of CNS involvement of ALL or with clinical signs or symptoms consistent with CNS involvement of ALL must undergo a lumbar puncture that is negative for CNS involvement of ALL
* Patients < 22 years of age must be willing to receive prophylactic intrathecal chemotherapy
* Must be registered on SWOG-9007 "Cytogenetic Studies in Leukemia Patients" (closed as of 07/01/2010)

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Serum creatinine ≤ 1.0 mg/dL OR glomerular filtration rate > 60 mL/min
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 1.5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment
* HIV-positive patients are eligible (at the discretion of the investigator) provided the following criteria are met:

  * No history of AIDS-defining conditions
  * CD4 cell count > 350/mm³
  * If on antiretroviral agents, must not include zidovudine or stavudine
  * Willing to receive prophylaxis for pneumocystis jirovecii pneumonia during study therapy (regardless of CD4 cell count) until the CD4 cell count is > 200/mm³ after completion of study treatment
* Prior malignancy (other than ALL) allowed provided it is in remission and there are no plans to treat the malignancy at the time of study registration
* No uncontrolled systemic fungal, bacterial, viral, or other infection, defined as exhibiting ongoing signs or symptoms related to the infection with no improvement despite appropriate antibiotics or other treatment
* No neuropathy (cranial, motor or sensory) ≥ grade 2

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Any number of prior therapies allowed
* More than 90 days since prior allogeneic bone marrow transplant (BMT)

  * No concurrent immunosuppression therapy for the treatment of graft-vs-host disease (GVHD)
  * No acute GVHD ≥ grade 2, moderate or severe limited chronic GVHD, or extensive chronic GVHD of any severity
* Prior autologous BMT allowed

  * No concurrent immunosuppression therapy for the treatment of GVHD
* More than 14 days since prior chemotherapy, investigational agents, or major surgery and recovered

  * Maintenance therapy with steroids, vincristine, and/or anti-metabolite agents, including but not limited to, mercaptopurine, thioguanine, and methotrexate allowed
  * Concurrent hydroxyurea to reduce WBC to a reasonable level (as deemed by the treating physician) allowed
* No prior clofarabine or epratuzumab
* No other concurrent cytotoxic therapy or investigational therapy
* No concurrent alternative medications (e.g., herbal or botanical medications for anticancer purposes)
* Concurrent participation on SWOG-S9910 "Leukemia Centralized Reference Laboratories and Tissue Repositories, Ancillary" allowed (closed as of 07/01/2010)

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Advani, MD, Study Chair — The Cleveland Clinic
Locations (81):
- United States (81):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - Stanford Cancer Center, Stanford, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Hematology-Oncology Clinic, Baton Rouge, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Saint Louis University Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Baylor University Medical Center - Houston, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - St. Luke's Texas Cancer Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Swedish Medical Center - Issaquah Campus, Issaquah, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Derived] Statler A, Othus M, Erba HP, Chauncey TR, Radich JP, Coutre S, Advani A, Nand S, Ravandi F, Mukherjee S, Sekeres MA. Comparable outcomes of patients eligible vs ineligible for SWOG leukemia studies. Blood. 2018 Jun 21;131(25):2782-2788. doi: 10.1182/blood-2018-01-826693. Epub 2018 Apr 4. PMID 29618479

RESULTS

PARTICIPANT FLOW:
Groups:
- Ara-C + Clofarabine + Epratuzumab: Ara-C 1 g/m2/d IV Days 1-5, clofarabine 40 mg/m2/d IV Days 2-6, epratuzumab 360 mg/m2/d IV Days 7, 14, 21, 28, acetaminophen 650 mg/d PO Days 7, 14, 21, 28, dephenhydramine 50 mg/d IV Days 7, 14, 21, 28, IT methotrexate 12 mg IT at least 1 wk apart during induction. 1 cycle=28 days. Maximum of one cycle.
Period: Overall Study
Arm/Group | Ara-C + Clofarabine + Epratuzumab
Started | 35
Eligible | 32
Eligible and Began Protocol Therapy | 31
Completed | 27
Not Completed | 8
Not completed — Death | 3
Not completed — Not protocol specified | 1
Not completed — Ineligible | 3
Not completed — Did not begin protocol therapy | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients who began protocol therapy were included in this analysis.
Arm/Group | Ara-C + Clofarabine + Epratuzumab
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 41 [21 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Secondary Outcome: Number of Patients With Grade 3 Through 5 Treatment-Related Adverse Events
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported. Any CTCAE 4.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Time Frame: Up to 5 years
Population: Eligible patients who received any treatment and were assessed for toxicity were included in the adverse event summaries.
Measure: Number; unit: Participants
Arm/Group | Ara-C + Clofarabine + Epratuzumab
Number analyzed (Participants) | 31
Participants
  Abdominal pain | 1
  Acute kidney injury | 1
  Alanine aminotransferase increased | 5
  Alkaline phosphatase increased | 1
  Anemia | 6
  Anorexia | 1
  Aspartate aminotransferase increased | 6
  Cardiac arrest | 2
  Catheter related infection | 2
  Diarrhea | 2
  Electrocardiogram QT corrected interval prolonged | 1
  Encephalopathy | 2
  Enterocolitis infectious | 2
  Febrile neutropenia | 17
  Gum infection | 1
  Hepatic failure | 1
  Hypercalcemia | 1
  Hyperglycemia | 1
  Hyperkalemia | 1
  Hypertension | 1
  Hypocalcemia | 1
  Hypokalemia | 1
  Hyponatremia | 1
  Hypophosphatemia | 1
  Hypotension | 2
  Hypoxia | 2
  Infections and infestations-Gram neg. bacteremia | 1
  Investigations - Bacteremia | 1
  Leukocytosis | 1
  Lung infection | 4
  Lymphocyte count decreased | 4
  Nervous system disorders - subdural hematoma | 1
  Neutrophil count decreased | 9
  Oral pain | 1
  Platelet count decreased | 12
  Respiratory failure | 1
  Sepsis | 4
  Tooth infection | 1
  Tumor lysis syndrome | 1
  Typhlitis | 2
  White blood cell decreased | 8

2. Primary Outcome: Complete Remission
Description: Complete remission (CR) is defined as: <5% marrow aspirate blasts. Blasts can be >=5% if the blasts are found to be myeloid and there is no evidence of lymphoblasts by flow cytometry or immunostaining. Neutrophils >= 1000/mcl; platelets >100,000/mcl; and no blasts in the peripheral blood. C1 Extramedullary disease status as defined in the protocol. Complete remission with incomplete platelet recovery (CRi) is same as CR but platelet count may be <=100,000/mcl and/or ANC may be <1,000/mcl.
Time Frame: After induction therapy was completed (1 or 2 months)
Population: Eligible patients who began protocol therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ara-C + Clofarabine + Epratuzumab
Number analyzed (Participants) | 31
percentage of participants | 52 [33 to 70]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Ara-C + Clofarabine + Epratuzumab
Serious Adverse Events (participants affected / at risk) | 15/31
Other Adverse Events (participants affected / at risk) | 27/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ara-C + Clofarabine + Epratuzumab (N=31)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Cardiac arrest (Cardiac disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 1
Typhlitis (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Catheter related infection (Infections and infestations) | 3
Enterocolitis infectious (Infections and infestations) | 1
Lung infection (Infections and infestations) | 3
Sepsis (Infections and infestations) | 4
Tooth infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Investigations - Other, specify (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Encephalopathy (Nervous system disorders) | 2
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Transient ischemic attacks (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ara-C + Clofarabine + Epratuzumab (N=31)
Anemia (Blood and lymphatic system disorders) | 10
Febrile neutropenia (Blood and lymphatic system disorders) | 13
Sinus tachycardia (Cardiac disorders) | 5
Ear pain (Ear and labyrinth disorders) | 2
Blurred vision (Eye disorders) | 2
Eye disorders - Other, specify (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 13
Dysphagia (Gastrointestinal disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 12
Chills (General disorders) | 5
Edema limbs (General disorders) | 4
Fatigue (General disorders) | 12
Fever (General disorders) | 4
Injection site reaction (General disorders) | 2
Localized edema (General disorders) | 2
Catheter related infection (Infections and infestations) | 2
Enterocolitis infectious (Infections and infestations) | 2
Gum infection (Infections and infestations) | 3
Lung infection (Infections and infestations) | 2
Papulopustular rash (Infections and infestations) | 2
Sepsis (Infections and infestations) | 4
Activated partial thromboplastin time prolonged (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 10
Alkaline phosphatase increased (Investigations) | 11
Aspartate aminotransferase increased (Investigations) | 12
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 2
INR increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 10
Platelet count decreased (Investigations) | 15
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 9
Anorexia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 14
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 12
Hypocalcemia (Metabolism and nutrition disorders) | 11
Hypoglycemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 8
Peripheral sensory neuropathy (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Hallucinations (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 5
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 7
Purpura (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Hematoma (Vascular disorders) | 3
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No